CLINICAL TRIAL: NCT01425697
Title: Randomized,Prospective Evaluation of 2% Chlorhexidine Gluconate Cloths to Reduce Surgical Site Infections in Cardiothoracic Surgery Patients
Brief Title: Eliminate Risk of Cardiac Surgical Site Events
Acronym: ERASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Sage Products, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Ackerman, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RSRB 25962
Record Dates: First submitted 2011-08-22; First posted 2011-08-30 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Surgical Site Infections
Keywords: Adult Cardiac surgery; Surgery site infections
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2% Chlorhexidine Gluconate cloths (Active Comparator): 2% Chlorhexidine Gluconate wipes will be used 12 hours prior to cardiac surgery and then again 3 hours prior to cardiac surgery
  Interventions: Other: 2% Chlorhexidine Gluconate cloths; Other: Standard of Care preoperative preparation.
- Standard of Care Preoperative Preparation (Other): Subject will receive standard of care preoperative preparation for the clinical site.
  Interventions: Other: 2% Chlorhexidine Gluconate cloths; Other: Standard of Care preoperative preparation.

INTERVENTIONS:
Other: 2% Chlorhexidine Gluconate cloths — 2% chlorhexidine Gluconate wipes will bw used 12 hours prior to cardiac surgery and then again 3 hours prior to cardiac surgery. Subjects will be randomized to either receive a preoperative phone call reminder or no phone call reminder.
Other: Standard of Care preoperative preparation. — Preoperative standard of care preparation utilized at the clinical site will be used. Subjects will be randomized to either receive a preoperative phone call reminder or no phone call reminder.

SUMMARY:
The purpose of the study is to see if using 2% Chlorhexidine cloths will reduce surgical site infections in patients having elective cardiac surgery.

DETAILED DESCRIPTION:
A randomized, prospective study utilizing 2% Chlorhexidine cloths to evaluate the product's effectiveness in reducing surgical site infections in elective cardiothoracic surgery patients. Sage 2% chlorhexidine cloths are approved by the Food and Drug Administration (FDA) for preparation of skin prior to surgery.

The study hypothesis is that the preoperative surgical preparation with 2% chlorhexidine cloths, which leaves chlorhexidine on the skin, will reduce surgical site infections by 50% as compared to current standard procedure.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiothoracic surgery patients > 18 years old.
* Informed consent obtained

Exclusion Criteria:

* Any current known allergies to chlorhexidine gluconate
* Currently taking any oral or topical antibiotics
* Any active skin rashes or breaks in the skin on areas to be treated with chlorhexidine gluconate
* A current active skin disease or inflammatory skin condition, known pre-existing skin infection, including contact dermatitis that is currently being treated with an antibiotic
* Any medical condition or use of any medications that in the opinion of the Principal Investigator preclude participation.
* Unwillingness or failure to fulfill requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 739 (Actual)
Dates: Start 2008-11; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Surgical site infections | Through 90 days post procedure
  Subjects will be assessed at 30 days and 90 days post operatively for any surgical site infection

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ackerman, DNS, Principal Investigator — University of Rochester
Locations (4):
- United States (4):
  - University of Kentucky, Lexington, Kentucky
  - The Valley Hospital, Ridgewood, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Robert Packer Hospital, Sayre, Pennsylvania

REFERENCES:
- [Result] DeBaun B. Evaluation of the antimicrobial properties of an alcohol-free 2% chlorhexidine gluconate (CHG) solution. Poster, accepted for presentation at: 2007 Association of perioperative registered nurses (AORN) Congress, Orlando, FL Mar 2007
- [Result] Ryder M. Improving Skin Antisepsis: 2% no-rinse CHG cloths improve antiseptic persistence on patient skin over 4% CHG rinse-off solution. Poster, accepted for presentation at:Association for Professionals in Infection Control and Epidemiology (APIC) June 2007
- [Result] Edmiston CE Jr, Seabrook GR, Johnson CP, Paulson DS, Beausoleil CM. Comparative of a new and innovative 2% chlorhexidine gluconate-impregnated cloth with 4% chlorhexidine gluconate as topical antiseptic for preparation of the skin prior to surgery. Am J Infect Control. 2007 Mar;35(2):89-96. doi: 10.1016/j.ajic.2006.06.012. PMID 17327187
- [Result] Edmiston C, Seabrook GR, Johnson CP, et al. Comparison of a new and innovative 2% chlorhexidine gluconate (CHG) impregnated preparation cloth with the standard 4% CHG surgical skin preparation. Poster, accepted for presentation at: 2007 Association of perioperative Registered Nurses (AORN) Congress, Orlando, FL Mar 2007.
- [Result] Eiselt D. Presurgical skin preparation with a novel 2% chlorhexidine gluconate (CHG) cloth leads to decrease in surgical site infection rates in orthopedic surgical patients. Poster accepted for presentation at: Association for Professionals in Infection Control and Epidemiology (APIC) June 2007.
- [Result] Rhee H, Harris B. Reducing surgical site infection: 2% CHG cloth reduces SSI rates by >70% difference resulting in a $154,869 cost avoidance. Poster accepted for presentation at: Virginians Improving Patient Care and Safety (VIPC&S) 7th Annual Conference.
- [Result] Berry AR, Watt B, Goldacre MJ, Thomson JW, McNair TJ. A comparison of the use of povidone-iodine and chlorhexidine in the prophylaxis of postoperative wound infection. J Hosp Infect. 1982 Mar;3(1):55-63. doi: 10.1016/0195-6701(82)90031-7. No abstract available. PMID 6177735